CLINICAL TRIAL: NCT02945735
Title: Gaze Contingent Feedback in Major Depressive Disorder
Brief Title: Gaze Contingent Feedback in Major Depressive Disorder (MDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor of Psychology and Neuroscience School of Psychological Sciences Sagol School of Neuroscience Tel Aviv University, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAUDEPI
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Depression, Unipolar; Depressive Disorder; Depressive Disorder, Major
Keywords: depression; cognitive bias modification; MDD; major depressive disorder; attention bias modification treatment
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- gaze-contingent (Experimental): Attention modification: participants will receive gaze-contingent feedback according to their viewing patterns
  Interventions: Behavioral: Attention Modification
- non-gaze contingent (Placebo Comparator): Participants will receive non-gaze-continent feedback unrelated to their viewing patterns
  Interventions: Behavioral: Attention Modification

INTERVENTIONS:
Behavioral: Attention Modification — Feedback according to participants' viewing patterns, in order to modify their attention.

SUMMARY:
The purpose of this study is to determine whether giving gaze-contingent feedback is an effective attention modification procedure, helping in the treatment of Major Depressive Disorder (MDD)

DETAILED DESCRIPTION:
The study examines giving depressive participants gaze-contingent feedback as a novel attention training procedure. Half of the participants will receive contingent feedback while the other half would receive non-contingent "placebo" feedback.

ELIGIBILITY:
Inclusion Criteria:

* A signed consent form
* Men and women between the ages of 18 and 65.
* Meeting a current diagnosis of Major Depressive Disorder (MDD) according to the DSM-IV
* MDD as the primary diagnosis: In cases of co-morbidity, MDD will be deemed as the most distressing and clinically significant condition among the co-morbid disorders
* Stable pharmaco-therapy: Participants receiving a pharmacological treatment who are taking a stable medication for at least 3 months before the beginning of the procedure.

Exclusion Criteria:

* Psychotic episode in the past or the present time.
* Co-morbidity with any neurological disorder (i.e., epilepsy, brain injury).
* Another psychotherapeutic treatment during the study.
* Usage of neuroleptic medication.
* Change in medication status during the study.
* Substantial usage of drugs or alcohol in the present time.
* Poor judgment capacity (i.e., children under 18 and special populations).
* High Risk of Suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-06 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline - Structured Interview for the Montgomery-Asberg Depression Rating Scale (SIGMA) | post treatment (1 week after treatment completion) and 3-month follow up
  The SIGMA is a ten-item diagnostic structured interview which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Each item is rated on scale ranging from 0 to 6 with a possible total score of 60, with regard to the passing week.

SECONDARY OUTCOMES:
Change from baseline - BDI-II - Beck Depression Inventory | post treatment (1 week after treatment completion) and 3-month follow up
  The BDI -II is a 21-question multiple-choice self-report inventory. Each item is rated on scale ranging from 0 to 3, Higher total scores indicate more severe depressive symptoms.

OTHER OUTCOMES:
changes in the Mini-International Neuropsychiatric Interview (M.I.N.I) diagnosis | approximately 20 min
  a structured diagnostic interview for DSM - IV and ICD-10 psychiatric disorders, which takes approximately 20 min to administer and is a valid and time-efficient alternative to the SCID-P and CIDI.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, Phd, Principal Investigator — Tel Aviv University
Locations (1):
- Tel-Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No